CLINICAL TRIAL: NCT05212090
Title: Study-Dependent Variability in Spinopelvic Parameters Among Patients Undergoing Total Hip Arthroplasty
Brief Title: Variability in Spinopelvic Parameters Among Patients Undergoing Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-011655
Record Dates: First submitted 2022-01-26; First posted 2022-01-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-THA (Other): Subjects will be receiving EOS imaging prior to Total Hip Arthroplasty (THA)
  Interventions: Diagnostic Test: EOS X-Ray
- Post-THA (Other): Subjects will be receiving EOS imaging after Total Hip Arthroplasty (THA)
  Interventions: Diagnostic Test: EOS X-Ray

INTERVENTIONS:
Diagnostic Test: EOS X-Ray — Repeated Anteroposterior (AP) Pelvis x-ray and Lateral Lumbar EOS x-ray

SUMMARY:
This research is being conducted to assess measurement correlations on different X-ray views on patients who have undergone or will undergo hip reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* 40 patients: 20 preoperative THA, 20 postoperative THA;
* Sex: 20 men, 20 women;
* Age: 20 patients ≥ 70 years, 10 patients 50-70 years, 10 patients 18-50 years.

Exclusion Criteria:

- Patients with lumbosacral hardware, contralateral THA.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Change in pelvic incidence (PI) | Baseline, 8 hours, 4 weeks
  Measured from EOS imaging and AP x-ray, reported in degrees
Change in symphysis to sacrococcygeal junction distance (PSCD) | Baseline, 8 hours, 4 weeks
  Measured from EOS imaging and AP x-ray, reported in millimeters (mm)
Change in pelvic tilt (PT) | Baseline, 8 hours, 4 weeks
  Measured from EOS imaging and AP x-ray, reported in degrees
Change in sacral slope (SS) | Baseline, 8 hours, 4 weeks
  Measured from EOS imaging and AP x-ray, reported in degrees
Change in lumbar lordosis (LL) | Baseline, 8 hours, 4 weeks
  Measured from EOS imaging and AP x-ray, reported in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abdel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials